CLINICAL TRIAL: NCT03612063
Title: Accuracy of Commercially Available Heart Rate Monitors in Athletes: A Prospective, Randomized Study
Brief Title: Accuracy of Commercially Available Heart Rate Monitors in Athletes
Acronym: HRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Milind Desai, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-800
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Heart Rate Monitors; Athletes Heart

STUDY DESIGN:
Intervention Model Description: The five heart rate monitors that will be assessed in this study include the Apple Watch Nike III, Fitbit Iconic, Garmin Vivosmart HR, TomTom Spark 3, and Polar H7 heart rate sensor. During testing, participants will wear two different wrist-worn heart rate monitors, the Polar H7 heart rate sensor, and will be connected to an ECG machine. Participants will be assigned, by chance to one of six groups:
  1. Fitbit Iconic HR and Garmin Vivosmart HR
  2. Fitbit Iconic HR and TomTom Spark 3
  3. Fitbit Iconic HR and Apple Watch III
  4. Apple Watch III and Garmin Vivosmart HR
  5. Apple Watch III and TomTom Spark 3
  6. Garmin Vivosmart HR and TomTom Spark 3
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Fitbit Iconic HR and Garmin Vivosmart HR (Experimental)
  Interventions: Device: Fitbit Iconic HR and Garmin Vivosmart HR
- Fitbit Iconic HR and TomTom Spark 3 (Experimental)
  Interventions: Device: Fitbit Iconic HR and TomTom Spark 3
- Garmin Vivosmart HR and TomTom Spark 3 (Experimental)
  Interventions: Device: Garmin Vivosmart HR and TomTom Spark 3
- Fitbit Iconic HR and Apple Watch III (Experimental)
  Interventions: Device: Fitbit Iconic HR and Apple Watch III
- Apple Watch III and Garmin Vivosmart HR (Experimental)
  Interventions: Device: Apple Watch III and Garmin Vivosmart HR
- Apple Watch III and TomTom Spark 3 (Experimental)
  Interventions: Device: Apple Watch III and TomTom Spark 3

INTERVENTIONS:
Device: Fitbit Iconic HR and Garmin Vivosmart HR — During testing, participants will wear two different wrist-worn heart rate monitors, the Polar H7 heart rate sensor, and will be connected to an ECG machine. Participants will be asked to perform a series of movements on a treadmill. Heart rate will be assessed under the following conditions:
  1. At rest
  2. 4 mph
  3. 5 mph
  4. 6 mph
  5. 7 mph
  6. 8 mph
  7. 9 mph
  8. Post-exercise 1 minute
  9. Post exercise 2 minutes
  Arms: Fitbit Iconic HR and Garmin Vivosmart HR
Device: Fitbit Iconic HR and TomTom Spark 3 — During testing, participants will wear two different wrist-worn heart rate monitors, the Polar H7 heart rate sensor, and will be connected to an ECG machine. Participants will be asked to perform a series of movements on a treadmill. Heart rate will be assessed under the following conditions:
  1. At rest
  2. 4 mph
  3. 5 mph
  4. 6 mph
  5. 7 mph
  6. 8 mph
  7. 9 mph
  8. Post-exercise 1 minute
  9. Post exercise 2 minutes
  Arms: Fitbit Iconic HR and TomTom Spark 3
Device: Garmin Vivosmart HR and TomTom Spark 3 — During testing, participants will wear two different wrist-worn heart rate monitors, the Polar H7 heart rate sensor, and will be connected to an ECG machine. Participants will be asked to perform a series of movements on a treadmill. Heart rate will be assessed under the following conditions:
  1. At rest
  2. 4 mph
  3. 5 mph
  4. 6 mph
  5. 7 mph
  6. 8 mph
  7. 9 mph
  8. Post-exercise 1 minute
  9. Post exercise 2 minutes
  Arms: Garmin Vivosmart HR and TomTom Spark 3
Device: Fitbit Iconic HR and Apple Watch III — During testing, participants will wear two different wrist-worn heart rate monitors, the Polar H7 heart rate sensor, and will be connected to an ECG machine. Participants will be asked to perform a series of movements on a treadmill. Heart rate will be assessed under the following conditions:
  1. At rest
  2. 4 mph
  3. 5 mph
  4. 6 mph
  5. 7 mph
  6. 8 mph
  7. 9 mph
  8. Post-exercise 1 minute
  9. Post exercise 2 minutes
  Arms: Fitbit Iconic HR and Apple Watch III
Device: Apple Watch III and Garmin Vivosmart HR — During testing, participants will wear two different wrist-worn heart rate monitors, the Polar H7 heart rate sensor, and will be connected to an ECG machine. Participants will be asked to perform a series of movements on a treadmill. Heart rate will be assessed under the following conditions:
  1. At rest
  2. 4 mph
  3. 5 mph
  4. 6 mph
  5. 7 mph
  6. 8 mph
  7. 9 mph
  8. Post-exercise 1 minute
  9. Post exercise 2 minutes
  Arms: Apple Watch III and Garmin Vivosmart HR
Device: Apple Watch III and TomTom Spark 3 — During testing, participants will wear two different wrist-worn heart rate monitors, the Polar H7 heart rate sensor, and will be connected to an ECG machine. Participants will be asked to perform a series of movements on a treadmill. Heart rate will be assessed under the following conditions:
  1. At rest
  2. 4 mph
  3. 5 mph
  4. 6 mph
  5. 7 mph
  6. 8 mph
  7. 9 mph
  8. Post-exercise 1 minute
  9. Post exercise 2 minutes
  Arms: Apple Watch III and TomTom Spark 3

SUMMARY:
The purpose of this research is to compare four different heart rate monitors (Apple Watch Nike III,Fitbit Iconic, Garmin Vivosmart HR, Tom Tom Spark 3) to an Electrocardiograph (ECG) machine to determine the accuracy of the devices. Over the last two decades, there has been a proliferation of commercially available heart rate monitors. Elite athletes often use heart rate measurements to monitor training and fitness levels. In response, fitness companies have offered a variety of heart rate monitors to the general public. Previously, chest strap monitors that measured electrical activity were mainly used to track heart rates. More recently, wrist-worn monitors that use an optical sensor (light) to measure heart rate have gained in popularity. While the accuracy of chest strap monitors has been studied, there is currently no data concerning the accuracy of wrist-worn heart rate monitors. Assessment of the monitors' accuracy is important for subjects who rely upon the heart rate measurements to guide their athletic activity.

DETAILED DESCRIPTION:
In 2018, worldwide sales of wearable fitness monitors are anticipated to exceed 110 million. Millions of consumers purchase fitness trackers that include heart rate monitors in order to help them to maintain their health and wellness. As popularity of these fitness devices grows, assessment and awareness of the accuracy of heart rate measurements becomes increasingly important.

In previous trials, the investigators assessed the accuracy of 4 wrist-worn HR monitors (Apple Watch, Fitbit Blaze, Garmin Forerunner 235, TomTom Spark Cardio) in healthy adult volunteers during various types of exercise. The investigators discovered that the accuracy varied with exercise type. With the treadmill, all devices were acceptable (rc =.88-.93) except the Fitbit Blaze (rc=.76). While biking, the Garmin and Apple Watch were acceptable (rc >.8). On the elliptical trainer without arm levers, only the Apple Watch provided accurate readings (rc=.94). None of the devices gave accurate readings for the elliptical trainer with arm levers (rc <.8). That study is now published.

Reviewers of the investigator's previous work raised an important question: how do commercial optical heart rate monitors perform when measuring heart rate in athletes performing at a high level of exertion? This study addresses that question.

The objective of this study is to evaluate the accuracy of four heart rate monitors in accomplished athletes (i.e. runners) performing at various levels of exertion, including a high level of exertion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients are able to run a mile in 7 minutes or less

Exclusion Criteria:

* Presence of a cardiac pacemaker
* Known chronic and persistent heart rhythm disorders
* Tattoos around the wrist or forearm area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
HR Monitor Assessment | 2 minutes of activity
  HR monitor values on each of the two wrist watches will be recorded along with the HR found on the Polar chest strap and ECG. In each running condition, heart rate will be assessed at 2 minutes of activity in order to ensure that a steady state heart rate has been achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Milind Desai, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No